CLINICAL TRIAL: NCT04613635
Title: Comparison of 2 Suture Materials for Closure of Ventral Defect At the Gastrojejunostomy in One-Anastomosis-Gastric Bypass / Mini-Gastric Bypass (OAGB / MGB): a Randomized Short Term Study with Monocrylic Spiral Knotless Tissue Control Device Vs. Traditional Polyglactin Multifilament Suture
Brief Title: Stratafix Vs. Vicryl OAGB / MGB Suture Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Franziskus Hospital (Other)
Collaborators: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Andreas Plamper, Assistant Principal Investigator, St. Franziskus Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191020
Record Dates: First submitted 2020-10-21; First posted 2020-11-03 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Morbid Obesity; Anastomotic Leak; Anastomotic Stenosis; Hemorrhage Postoperative
Keywords: Mini-Gastric Bypass; One Anastomosis Gastric Bypass; Gastroenteral Anastomosis; MGB; OAGB
MeSH Terms: conditions — Obesity, Morbid; Anastomotic Leak; Postoperative Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stratafix (Experimental)
  Interventions: Device: Stratafix
- Vicryl (Active Comparator)
  Interventions: Device: Vicryl

INTERVENTIONS:
Device: Stratafix — Closure of ventral defect of the otherwise stapled gastrojejunal anastomosis with Stratafix USP (United States Pharmacopoe) 2-0 thread
  Other Names: monocrylic spiral knotless tissue control device
  Arms: Stratafix
Device: Vicryl — Closure of ventral defect of the otherwise stapled gastrojejunal anastomosis with Vicryl USP 2-0 thread
  Other Names: traditional polyglactin multifilament suture
  Arms: Vicryl

SUMMARY:
To compare shorttime (6 months) results of two competitive suture materials with regard to time demanded to perform the concerned surgical step and secondary to study anastomotic site safety and complications like leakage and hemorrhage as well as development of anastomotic strictures. Evaluation of cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* adult patients selected for primary Mini-Gastric bypass to treat obesity (BMI>30)
* laparoscopic access feasable (intention to treat laparoscopically)
* failed conservative treatment (accepted by health insurance companies)
* relevant co-morbidities in cases with BMI <40
* age 18 years or elder

Exclusion Criteria:

* severe language problems
* revisional or redo-procedures
* operation intended as open procedure(extensive previous surgeries),
* operation performed under corticoid-medication
* operation performed under full-dose anticoagulants
* operation performed by another surgeon than one of the 3 experienced MGB-surgeons of the Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Closure of gastrojejunostomy | The assessment of this surgical step will be completed during the operation.
  time needed to perform this specific surgical step, i.e. the ventral defect closure of the (otherwise stapled) gastrojejunostomy

SECONDARY OUTCOMES:
anastomotic site perioperative morbidity | 6 months
  Number of participants with hemorrhage, leakage or symptomatic strictures requiring further diagnostic or therapeutic measurements
other anastomosis- related morbidity | 6 months
  Number of participants with marginal ulcer or anastomotic stricture needing further diagnostic and/or interventions
economical factors | 6 months
  costs of treatment in case the above mentioned complications occur and require intervention

CONTACTS AND LOCATIONS:
Locations (1):
- St. Franziskus-Hospital, Cologne, Germany

REFERENCES:
- [Background] Lee WJ, Ser KH, Lee YC, Tsou JJ, Chen SC, Chen JC. Laparoscopic Roux-en-Y vs. mini-gastric bypass for the treatment of morbid obesity: a 10-year experience. Obes Surg. 2012 Dec;22(12):1827-34. doi: 10.1007/s11695-012-0726-9. PMID 23011462
- [Background] Rutledge R, Walsh TR. Continued excellent results with the mini-gastric bypass: six-year study in 2,410 patients. Obes Surg. 2005 Oct;15(9):1304-8. doi: 10.1381/096089205774512663. PMID 16259892
- [Background] Kular KS, Manchanda N, Rutledge R. A 6-year experience with 1,054 mini-gastric bypasses-first study from Indian subcontinent. Obes Surg. 2014 Sep;24(9):1430-5. doi: 10.1007/s11695-014-1220-3. PMID 24682767
- [Background] Chevallier JM, Arman GA, Guenzi M, Rau C, Bruzzi M, Beaupel N, Zinzindohoue F, Berger A. One thousand single anastomosis (omega loop) gastric bypasses to treat morbid obesity in a 7-year period: outcomes show few complications and good efficacy. Obes Surg. 2015 Jun;25(6):951-8. doi: 10.1007/s11695-014-1552-z. PMID 25585612
- [Background] Noun R, Skaff J, Riachi E, Daher R, Antoun NA, Nasr M. One thousand consecutive mini-gastric bypass: short- and long-term outcome. Obes Surg. 2012 May;22(5):697-703. doi: 10.1007/s11695-012-0618-z. PMID 22411569
- [Background] Musella M, Susa A, Greco F, De Luca M, Manno E, Di Stefano C, Milone M, Bonfanti R, Segato G, Antonino A, Piazza L. The laparoscopic mini-gastric bypass: the Italian experience: outcomes from 974 consecutive cases in a multicenter review. Surg Endosc. 2014 Jan;28(1):156-63. doi: 10.1007/s00464-013-3141-y. Epub 2013 Aug 28. PMID 23982648
- [Background] Taha O, Abdelaal M, Abozeid M, Askalany A, Alaa M. Outcomes of Omega Loop Gastric Bypass, 6-Years Experience of 1520 Cases. Obes Surg. 2017 Aug;27(8):1952-1960. doi: 10.1007/s11695-017-2623-8. PMID 28303503
- [Background] Carbajo MA, Luque-de-Leon E, Jimenez JM, Ortiz-de-Solorzano J, Perez-Miranda M, Castro-Alija MJ. Laparoscopic One-Anastomosis Gastric Bypass: Technique, Results, and Long-Term Follow-Up in 1200 Patients. Obes Surg. 2017 May;27(5):1153-1167. doi: 10.1007/s11695-016-2428-1. PMID 27783366
- [Background] Lee WJ, Wang W, Lee YC, Huang MT, Ser KH, Chen JC. Laparoscopic mini-gastric bypass: experience with tailored bypass limb according to body weight. Obes Surg. 2008 Mar;18(3):294-9. doi: 10.1007/s11695-007-9367-9. Epub 2008 Jan 12. PMID 18193178
- [Background] Skroubis G, Sakellaropoulos G, Pouggouras K, Mead N, Nikiforidis G, Kalfarentzos F. Comparison of nutritional deficiencies after Roux-en-Y gastric bypass and after biliopancreatic diversion with Roux-en-Y gastric bypass. Obes Surg. 2002 Aug;12(4):551-8. doi: 10.1381/096089202762252334. PMID 12194550